CLINICAL TRIAL: NCT06337110
Title: Interventional, Open-label, Single-dose Trial Investigating the Absorption, Metabolism, and Excretion (AME) of Lu AF28996 Following a Single Oral Dosing of 14C-Lu AF28996 to Healthy Men
Brief Title: A Study Investigating the Movement of Lu AF28996 Into, Through, and Out of the Body of Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20436A
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lu AF28996 (Experimental): Participants will receive a single oral dose of Lu AF28996.
  Interventions: Drug: Lu AF28996

INTERVENTIONS:
Drug: Lu AF28996 — Oral solution containing radiolabelled [14C]-Lu AF28996.

SUMMARY:
The main goal of this study is to learn about how Lu AF28996 moves into, through, and out of the body after a single dose is given to healthy male participants.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant has a Body Mass Index (BMI) >=18.5 and <=30 kilograms per square meter (kg/m^2) and body weight ≥60 kg at the Screening Visit and at the Baseline Visit.
* The participant has a resting supine pulse >=50 and <=100 beats per minute (bpm) at the Screening Visit and at the Baseline Visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, a neurological examination, vital signs, an electrocardiogram (ECG), and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Key Exclusion Criteria:

* The participant has participated in a clinical trial <30 days prior to the Screening Visit.
* The participant has taken any investigational medicinal product <3 months or <5 half-lives of that product, whichever is longest, prior to the first dose of investigational medicinal product (IMP).
* Participants with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.

Other protocol-defined criteria apply.

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Total Recovery of the Administered Radiolabelled Drug-related Material (Percentage of Dose in Urine and Faeces) | From baseline (Day -1) up to 23 days post-dose
AUC0-infinity: Area Under the Plasma Concentration Curve of Radiolabelled Drug-related Material from Zero to Infinity | From date of dosing (Day 1) up to 23 days post-dose
Cmax: Maximum Observed Plasma Concentration of Radiolabelled Drug-related Material | From date of dosing (Day 1) up to 23 days post-dose
Tmax: Nominal Time Corresponding to the Occurrence of Cmax of Radiolabelled Drug-related Material | From date of dosing (Day 1) up to 23 days post-dose
T½: Apparent Elimination Half-life of Radiolabelled Drug-related Material | From date of dosing (Day 1) up to 23 days post-dose
AUC0-infinity of Lu AF28996 | From date of dosing (Day 1) up to 23 days post-dose
Cmax of Lu AF28996 | From date of dosing (Day 1) up to 23 days post-dose
Tmax of Lu AF28996 | From date of dosing (Day 1) up to 23 days post-dose
T½ of Lu AF28996 | From date of dosing (Day 1) up to 23 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea Clinical Research Unit Ltd, Leeds, United Kingdom